CLINICAL TRIAL: NCT05653310
Title: Pharmacodynamics, Pharmacogenetics, Clinical Efficacy and Safety of Tradipitant for Functional Dyspepsia
Brief Title: Tradipitant for Functional Dyspepsia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Xiao Jing (Iris) Wang (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Xiao Jing (Iris) Wang, Regulatory Sponsor and Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 21-012527
Record Dates: First submitted 2022-04-29; First posted 2022-12-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Functional Dyspepsia
Keywords: tradipitant; NK-1 antagonist; neurokinin 1 receptor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tradipitant (Experimental): Oral Capsule
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator): Oral Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tradipitant — Tradipitant Capsule
  Arms: Tradipitant
Drug: Placebo — Placebo Capsule
  Arms: Placebo

SUMMARY:
To evaluate the effects of tradipitant relative to placebo on gastric motor functions, satiation, and postprandial symptoms in patients with functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent
* Body Mass Index (BMI) of 18-35 kg/m2
* Absence of other diseases which could interfere with interpretation of study results

Exclusion Criteria:

* Current H. pylori infection
* Pregnancy or nursing
* Recent history of Alcohol Use Disorder or Substance Use Disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Accommodation gastric volumes measured by single photon emission computed tomography (SPECT) | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Jing (Iris) Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials